CLINICAL TRIAL: NCT03270813
Title: RAGE-Control: Teaching Emotional Self-regulation Through Videogame Play
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Academy of Child Adolescent Psychiatry. (Other); Harvard University (Other)
Responsible Party: Principal Investigator, Carrie Vaudreuil, Assistant in Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015P000901
Record Dates: First submitted 2017-06-28; First posted 2017-09-01 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Anger; Aggression
Keywords: Child; Adolescent
MeSH Terms: conditions — Aggression | interventions — Relaxation Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RAGE-Control (Experimental): There are 6 research intervention sessions, which will involve Relaxation training plus RAGE-Control. The first session includes a 30-minute lesson on the relationship between physiological arousal and anger, introduction to the RAGE-Control videogame and 15 minutes of videogame play. The next 5 sessions include a 10-minute check in about symptoms and functioning, a brief presentation of a relaxation skill, and 15 minutes of videogame play.
  Interventions: Behavioral: Relaxation training plus RAGE-Control
- Sham videogame (Sham Comparator): There are 6 research intervention sessions, which will involve Relaxation training plus Sham videogame. The first session includes a 30-minute lesson on the relationship between physiological arousal and anger, an introduction to the Sham videogame and 15 minutes of videogame play. The next 5 sessions include a 10-minute check in about symptoms and functioning, a brief presentation of a relaxation skill, and 15 minutes of videogame play.
  Interventions: Behavioral: Relaxation training plus Sham Videogame

INTERVENTIONS:
Behavioral: Relaxation training plus RAGE-Control — RAGE-Control is a biofeedback videogame in which players shoot at enemies while avoiding allies. The player's baseline heart rate is taken before the game and entered into the computer. During the game, the player wears a heart rate monitor, and if the player's heart rate rises above baseline, they are unable to shoot. The player must use relaxation skills to decrease their heart rate below the baseline before they can resume play. Participants will undergo relaxation training during each of 6 sessions, and then practice the skills they learned while playing the RAGE-Control videogame.
  Other Names: RAGE-Control
  Arms: RAGE-Control
Behavioral: Relaxation training plus Sham Videogame — The Sham videogame is a videogame in which players shoot at enemies while avoiding allies. The player wears a heart rate monitor during the game, but the heart rate does not affect the functioning of the game in any way. Participants will undergo relaxation training during each of 6 sessions, and then practice the skills they learned while playing the Sham videogame.
  Other Names: Sham Videogame
  Arms: Sham videogame

SUMMARY:
The purpose of this study is to evaluate the use of Regulate and Gain Emotional Control (RAGE-Control), a biofeedback video game, in combination with brief instruction in relaxation skills as an intervention for symptoms of anger and aggression in children and adolescents. Half of the research participants will learn relaxation techniques and practice them using the RAGE-Control videogame. The other half of the participants will learn relaxation techniques and play a similar videogame without the biofeedback component. The investigators hypothesize that participants in the RAGE-Control group will show a greater reduction in symptoms of anger and aggression than those in the non-RAGE-Control group.

DETAILED DESCRIPTION:
Experiencing mild anger and aggression in frustrating situations is typical in childhood; however, over time most children develop the capacity to regulate their anger in emotionally provoking situations. Those who continue to struggle with emotional and behavioral regulation are at heightened risk for social isolation, delinquency, substance abuse, and academic problems later in life. Moreover, adults who were aggressive as children experience poor physical and mental health, and may find limited career opportunities.

Although anger regulation is a common and clinically significant psychiatric concern for children and adolescents, effective treatment options are limited. As a result, clinicians increasingly rely on psychotropic medications to blunt anger. Psychotropic medications can reduce anger and aggression in the short term, but they fail in the long-term goal of teaching self-regulation, and carry the risk of serious side-effects, including obesity, metabolic syndrome, and type II diabetes. However, engaging youth with anger issues in therapeutic treatments can be difficult, with high rates of attrition. These difficulties underline the need for innovative treatments that can effectively engage patients and enhance their ability to control their emotions and behaviors.

In response to this need, clinicians at Boston Children's Hospital developed Regulate and Gain Emotional Control (RAGE-Control), a therapeutic videogame that requires players to maintain low levels of physiologic arousal while rapidly reacting to incoming stimuli and inhibiting erroneous responses. It was initially designed for use with Cognitive Behavioral Therapy (CBT) to motivate children to remain engaged in therapy, and to foster the learning, practice, and generalization of self-regulation skills in the midst of frustrating or anger provoking situations. Pilot data from an open label trial of RAGE-Control on a pediatric psychiatric inpatient unit demonstrated improvement in patient self-reported anger and aggression after 5 sessions of CBT with RAGE-Control, when compared with a treatment as usual group. A subsequent outpatient randomized controlled trial comparing CBT with RAGE-Control to CBT with a sham videogame demonstrated that patients who participated in the RAGE-Control intervention had significantly greater improvements in overt aggression and oppositionality, parental stress, and family atmosphere. The participants in the RAGE-Control group also had fewer drop outs, and twice as many treatment responders as the participants in the control arm.

ELIGIBILITY:
Inclusion Criteria:

* Problems with anger and/or aggression
* Score of at least 4/10 on phone screen with parents measuring anger and aggression

Exclusion Criteria:

* Changes in dosing of psychotropic medications within the 8 weeks prior to the start of the study, or anticipated medication changes during the study.
* Starting therapy within the 8 weeks prior to starting the study, or anticipated new therapy beginning during the study.
* Actively participating in any type of Cognitive Behavioral Therapy for less than 12 weeks and/or attending Cognitive Behavioral Therapy weekly or more.
* Intellectual disability (IQ < 80)
* Suicidal ideation
* Homicidal ideation
* Psychosis/meets criteria for psychotic disorder

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-03 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Impressions Global Rating of Improvement (CGI-I) | Up to 3 months post-intervention
  Assesses improvement post treatment, with scores ranging from 1 (very much improved) to 7 (very much worse).

SECONDARY OUTCOMES:
Clinical Global Impressions Severity of Illness (CGI-S) | Up to 3 months post intervention
  Assess overall burden of illness on a scale from 1 (normal, not ill) to 7 (very severely ill).
State Trait Anger Expression Inventory for Children and Adolescents (STAXI-CA) | Baseline, 2 weeks post treatment, 3 months post treatment
  35 item self-report scale that assesses state anger, trait anger and expression of anger.
Multidimensional Adolescent Satisfaction Scale (MASS) | 2 weeks post treatment, 3 months post treatment
  Measures patient satisfaction with the intervention
Modified Overt Aggression Scale (MOAS) | Baseline, 2 weeks post treatment, 3 months post treatment
  Records the severity of 4 types of aggression: verbal, against property, physical, and against self.
Difficulties in Emotion Regulation Scale (DERS) | Baseline, 2 weeks post treatment, 3 months post treatment
  36-item, self-report questionnaire designed to assess multiple aspects of emotion dysregulation. For patients age 10 and older only.
Difficulties in Emotion Regulation Scale - impulse control difficulties | Up to 3 months post intervention
  6 items of the DERS specifically designed to assess impulse control difficulties. For patients age 10 and older only.
Child Behavior Checklist (CBCL) 6-18 | Baseline, 2 weeks post treatment, 3 months post treatment
  Empirically based checklist of social competence and behavioral problems, filled out by parents based on recent behavior.
Heart rate | Weekly for 6 weeks
  The computer will record each participant's heart rate while they play the videogame.
Emotion Regulation Checklist (ERC) | Up to 3 months post intervention
  24 item parent-report questionnaire regarding a child's ability to assess emotion regulation in the past 1 week.

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Vaudreuil, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kahn J, Ducharme P, Rotenberg A, Gonzalez-Heydrich J. "RAGE-Control": A Game to Build Emotional Strength. Games Health J. 2013 Feb;2(1):53-7. doi: 10.1089/g4h.2013.0007. PMID 26196556
- [Background] Kahn J, Ducharme P, Travers B, Gonzalez-Heydrich J. RAGE Control: Regulate and Gain Emotional Control. Stud Health Technol Inform. 2009;149:335-43. PMID 19745492
- [Background] Ducharme P., Wharff E., Kahn J., Hutchinson E., & Logan G. Augmenting anger control therapy with a videogame requiring emotional control: A pilot study on an inpatient psychiatric unit. Adolescent Psychiatry, 2012; 2(4), 323-332.
- [Derived] Vaudreuil C, Abel MR, Barnett Y, DiSalvo M, Hirshfeld-Becker DR. A Pilot Controlled Trial of Relaxation Training Combined with a Video Game Reinforcing Emotional Regulation to Improve Anger Management in Children and Adolescents. Res Child Adolesc Psychopathol. 2024 Dec;52(12):1847-1859. doi: 10.1007/s10802-024-01259-w. Epub 2024 Oct 23. PMID 39441503